CLINICAL TRIAL: NCT03087409
Title: High-dose Chemotherapy With Hematopoietic Stem-cell Rescue for High-risk Breast Cancer: Long-term Follow-up of a Randomized Phase III Study
Brief Title: High-dose Chemotherapy With Hematopoietic Stem-cell Rescue for High-risk Breast Cancer: Long-term Follow-up
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 201600539
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Collection of follow-up data from the original trial patient cohort.

DETAILED DESCRIPTION:
Collection of follow-up data from the original trial patient cohort by means of structured patient file abstraction, a questionnaire to the general practitioner, and registry consultations.

ELIGIBILITY:
Inclusion Criteria:

* Enrolment in the original trial.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage II or III breast cancer involving ≥ 4 axillary lymph nodes, who have been treated with adjuvant chemotherapy with or without intensification and hematopoietic stem-cell rescue.
Sampling Method: Non-Probability Sample
Enrollment: 885 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Overall survival according to the definition and analysis plan of the original study
Relapse-free survival | 2 years
  Relapse-free survival according to the definition and analysis plan of the original study

SECONDARY OUTCOMES:
Incidence of cardiovascular events | 2 years
Incidence of malignancies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: J A Gietema, MD, PhD, Principal Investigator — University Medical Center Groningen; G Sonke, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (10):
- Netherlands (10):
  - Academic Medical Center, Amsterdam
  - The Netherlands Cancer Institute, Amsterdam
  - VU University Medical Center, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodenhuis S, Bontenbal M, Beex LV, Wagstaff J, Richel DJ, Nooij MA, Voest EE, Hupperets P, van Tinteren H, Peterse HL, TenVergert EM, de Vries EG; Netherlands Working Party on Autologous Transplantation in Solid Tumors. High-dose chemotherapy with hematopoietic stem-cell rescue for high-risk breast cancer. N Engl J Med. 2003 Jul 3;349(1):7-16. doi: 10.1056/NEJMoa022794. PMID 12840087
- [Derived] Steenbruggen TG, Steggink LC, Seynaeve CM, van der Hoeven JJM, Hooning MJ, Jager A, Konings IR, Kroep JR, Smit WM, Tjan-Heijnen VCG, van der Wall E, Bins AD, Linn SC, Schaapveld M, Jacobse JN, van Leeuwen FE, Schroder CP, van Tinteren H, de Vries EGE, Sonke GS, Gietema JA. High-Dose Chemotherapy With Hematopoietic Stem Cell Transplant in Patients With High-Risk Breast Cancer and 4 or More Involved Axillary Lymph Nodes: 20-Year Follow-up of a Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Apr 1;6(4):528-534. doi: 10.1001/jamaoncol.2019.6276. PMID 31999296